CLINICAL TRIAL: NCT02826161
Title: A Phase III Randomized, Open-Label Clinical Trial of BBI-608 Plus Weekly Paclitaxel Versus Weekly Paclitaxel Alone in Patients With Advanced, Previously Treated, Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of Napabucasin (BBI-608) Plus Weekly Paclitaxel Versus Weekly Paclitaxel Alone in Patients With Advanced, Previously Treated, Non-Squamous Non-Small Cell Lung Cancer
Acronym: CanStem43L
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change of treatment landscape and evolving standard of care
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanStem43L
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Neoplasms; Neoplasms by Site; Lung Neoplasms; Thoracic Neoplasms; Respiratory Tract Neoplasms; Bronchial Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasms by Site; Lung Neoplasms; Thoracic Neoplasms; Respiratory Tract Neoplasms; Bronchial Neoplasms | interventions — napabucasin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Napabucasin plus Weekly Paclitaxel (Experimental): Patients randomized to this arm will receive napabucasin administered orally, twice daily in combination with paclitaxel administered intravenously, once weekly, on 3 of every 4 weeks.
  Interventions: Drug: Napabucasin; Drug: Paclitaxel
- Weekly Paclitaxel (Active Comparator): Patients randomized to this arm will receive weekly paclitaxel alone administered intravenously, once weekly, on 3 of every 4 weeks.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Napabucasin — Napabucasin will be administered in continuous 28-day cycles. The starting dose of napabucasin is 240 mg twice daily (480 mg total daily dose) with approximately 12 hours between each dose. Napabucasin should be taken with fluids either 1 hour prior to a meal or 2 hours after a meal.
  Other Names: BBI-608; BBI608; BB608
  Arms: Napabucasin plus Weekly Paclitaxel
Drug: Paclitaxel — Paclitaxel will be administered intravenously, once weekly, via one-hour infusion at a starting dose-level of 80 mg/m^2 body surface area. The weekly paclitaxel infusion will be given during 3 out of every 4 weeks, on days 1, 8, and 15 of each 28-day study cycle.

SUMMARY:
This is an international, multi-center, prospective, randomized, open-label Phase 3 clinical trial of the cancer stemness inhibitor napabucasin administered with weekly paclitaxel versus weekly paclitaxel alone in patients with advanced non-squamous non-small cell lung cancer who have disease progression following systemic treatment with a platinum-based combination regimen in the metastatic setting, who have received treatment with an immune checkpoint inhibitor if a candidate, additional approved therapies, and for whom weekly paclitaxel is an acceptable treatment option.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have histologically or cytologically confirmed non-squamous NSCLC.
* Must have progressed following treatment with platinum-based combination chemotherapy for metastatic disease, and patients with an EGFR or ALK/ROS1 genetic aberration must have received appropriately targeted treatment.
* Must have received either nivolumab or pembrolizumab or a different IND-approved anti-PD1 or anti-PD-L1 therapy, unless medically contraindicated
* Weekly paclitaxel must be an acceptable treatment option
* Must submit tumor tissue for correlative analyses
* Women of child-bearing potential and partners of women of child-bearing potential must take measures to avoid pregnancy while receiving and for a period of time following protocol therapy
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, adequate organ function, and a life expectancy of ≥ 3 months

Key Exclusion Criteria:

* Has squamous NSCLC
* Has received prior systemic treatment with a taxane for advanced/metastatic disease
* Has received systemic anti-cancer therapy within the 14 days prior to randomization
* Has received radiotherapy within the 28 days prior to randomization, with the exception of palliative radiotherapy to focal lesions for pain or other symptom control
* Has brain metastases with evolving neurologic symptoms or a steroid requirement.
* Has had major surgery requiring general anesthesia and/or mechanical ventilation within the 28 days prior to randomization
* Has a corrected QT interval (QTc) > 470 ms or has an electrocardiogram (ECG) with a new abnormal finding that is clinically significant
* Has peripheral neuropathy ≥ Grade 2 (NCI-CTCAE)
* Refuses to complete quality of life questionnaires either alone or with assistance from study staff despite adequate fluency
* Has an intercurrent (non-malignant) chronic medical or psychiatric illness or condition(s) not optimally controlled and carrying a moderate to high risk of interfering with protocol therapy administration or compliance with required procedures, in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Beverly Hills, California
  - Santa Rosa, California
  - Aventura, Florida
  - Gettysburg, Pennsylvania
  - Arlington, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Napabucasin Plus Paclitaxel: All participants were randomized to receive napabucasin (BBI-608) 240 mg administered orally, twice daily (480 mg total in a day) plus Paclitaxel 80 mg/m2 IV; once weekly ( three out of every four weeks)
- Paclitaxel Only: All participants were randomized to receive Paclitaxel 80 mg/m2 IV, once weekly ( three out of every four weeks)
Period: Overall Study
Arm/Group | Napabucasin Plus Paclitaxel | Paclitaxel Only
Started | 1 | 3
Discontinued Due to Treatment Related AE | 1 | 0
Discontinued Due to Death | 0 | 1
Discontinued Due to Patient Withdrawal | 0 | 1
Discontinued Due to Withdrawal of ICF From Further FU | 1 | 1
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Napabucasin Plus Paclitaxel: All participants randomized to receive napabucasin (BBI-608) 240 mg twice daily administered orally, twice daily (480 mg total in a day) plus Paclitaxel 80 mg/m2 IV; once weekly ( three out of every four weeks)
- Paclitaxel Only: All participants randomized to receive Paclitaxel 80 mg/m2 IV, once weekly ( three out of every four weeks)
- Total: Total of all reporting groups
Arm/Group | Napabucasin Plus Paclitaxel | Paclitaxel Only | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To assess the effect of napabucasin plus weekly paclitaxel versus weekly paclitaxel on the Overall Survival of patients with previously treated advanced, non-squamous non-small cell lung cancer.
Time Frame: 36 months
Population: The study was terminated early by the sponsor after 4 patients were randomized (3 to the control arm and 1 to receive napabucasin). Due to the small sample size, no data summaries were performed and there is no analysis for statistical interference.
Groups:
- All Participants: All participants were randomized to receive either napabucasin (BBI-608) 240 mg twice daily administered orally, twice daily (480 mg total in a day) plus Paclitaxel 80 mg/m2 IV; weekly ( three out of every four weeks) or, Paclitaxel 80 mg/m2 IV, weekly ( three out of every four weeks)
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly paclitaxel versus weekly paclitaxel on the Overall Survival of patients with previously treated advanced, non-squamous non-small cell lung cancer in biomarker positive patients. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival
Description: To assess the effect of napabucasin plus weekly paclitaxel versus weekly paclitaxel on the Progression Free Survival (PFS) of patients with previously treated advanced, non-squamous non-small cell lung cancer. PFS is defined as the time from randomization to the first objective documentation of disease progression or death due to any cause.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly paclitaxel versus weekly paclitaxel on the Progression Free Survival (PFS) of patients with previously treated advanced, non-squamous non-small cell lung cancer in biomarker positive patients. PFS is defined as the time from randomization to the first objective documentation of disease progression or death due to any cause. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Disease Control Rate in Biomarker Positive Patients
Description: To assess the effect of napabucasin plus weekly paclitaxel versus weekly paclitaxel on the Disease Control Rate (DCR) of patients with previously treated advanced, non-squamous non-small cell lung cancer. DCR is defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1. This biomarker-positive sub-population is defined as those patients with phospho-STAT3 based on immunohistochemical (IHC) staining of Formalin Fixed Paraffin Embedded (FFPE) tumor tissue.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Quality of Life (QoL)
Description: QoL will be measured using the European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC-QLQ-C30) in patients with previously treated advanced, non-squamous non-small cell lung cancer with napabucasin plus weekly paclitaxel versus weekly paclitaxel.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Disease Control Rate
Description: To assess the effect of napabucasin plus weekly paclitaxel versus weekly paclitaxel on the Disease Control Rate (DCR) of patients with previously treated advanced, non-squamous non-small cell lung cancer. DCR is defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Patients With Adverse Events
Description: All patients who have received at least one dose of napabucasin will be included in the safety analysis according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.0. The incidence of adverse events will be summarized by type of adverse event and severity.
Time Frame: 36 months
Population: as for outcome 1
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The safety documentation and reporting begins with completion of the informed consent and extends until 30 days following the last dose of the protocol therapy, the total period is 36 months
Groups:
- Napabucasin+Paclitaxel: All participants part of the safety population ( those who received at least 1 dose of study drug napabucasin).
- Paclitaxel Only: All participants part of the safety population ( those who received at least 1 dose of paclitaxel).
Arm/Group | Napabucasin+Paclitaxel | Paclitaxel Only
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin+Paclitaxel (N=1) | Paclitaxel Only (N=2)
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Costipation (Gastrointestinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Edema Lower Legs (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
On 12 June 2017 the sponsor notified study investigator that the study was terminated because of the rapidly evolving standard of care for patients with NSCLC. At the time of the termination, there were only 4 patients randomized (3 to the control arm and 1 to the napabucasin arm). Due to the small sample size, neither safety or efficacy data were analyzed or summarized for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before submission for publication or presentation, Institution and/or Investigator shall allow Sponsor not less than sixty ( 60) days to review any manuscript and not less than thirty ( 30) days to review any poster presentation, abstract or any other written or oral material which describes or discloses the study results. If Sponsor requests in writing, institution and/or Investigator shall withhold any publication or presentation for an additional sixty ( 60) days.

DOCUMENTS (2):
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT02826161/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT02826161/SAP_001.pdf